CLINICAL TRIAL: NCT02374281
Title: Autonomic Nervous System Reactivity of the Newborn After a Nociceptive Stress: Interest of Sucrose and Non-nutritive Sucking : A Controlled Randomized Single-center Study.
Brief Title: Autonomic Nervous System Reactivity of the Newborn After a Nociceptive Stress: Interest of Sucrose and Non-nutritive Sucking
Acronym: BBSUCROSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1308143; 2013-005043-86 (EudraCT Number)
Record Dates: First submitted 2015-02-10; First posted 2015-02-27 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Newborn; Neonatal Screening
Keywords: Newborn; Neonatal Screening; Autonomic Nervous System; Pain; non-nutritive sucking; sucrose administration; nociceptive action; Electro acoustical characteristics of crying
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucose sucking (Experimental): The newborn will receive one minute before the painful care either a compress with sucrose.
  The puncture made in the veins of the back of the hand, will be performed only once per patient per test.
  Glucose 30% by oral route (1 ml).
  Interventions: Drug: Glucose sucking
- Water sucking (Active Comparator): The newborn will receive one minute before the painful care either a compress with water.
  The puncture made in the veins of the back of the hand, will be performed only once per patient per test.
  Sterile water by oral route (1 ml).
  Interventions: Drug: Water sucking
- No sucking (Placebo Comparator): The puncture made in the veins of the back of the hand, will be performed only once per patient per test.
  Interventions: Other: No sucking

INTERVENTIONS:
Drug: Glucose sucking
  Other Names: Glucose PROAMP 30%, Laboratoires AGUETTANT
  Arms: Glucose sucking
Drug: Water sucking
  Other Names: Eau ppi, BRAUN
  Arms: Water sucking
Other: No sucking
  Arms: No sucking

SUMMARY:
The management of the pain is a constant care concern in neonatal and maternity units. Many studies show an interest in the use of sugar solutions to reduce nociception during painful events in infants. However, these studies are based mainly on behavioral observation of the newborn but intrinsic mechanisms of analgesic power are not clearly understood for sucrose solutions.

Our hypothesis is that the analgesic mechanism of sucrose solutions in infants involves a subcortical reactivity notably by action via the brain stem. To explore the intensity of pain and evaluate the subcortical activity, we will use 1) the analysis of heart rate variability (frequency indices whose HFnu) as a peripheral witness of subcortical functioning of the autonomic nervous system 2) electroacoustic analysis of the intensity of crying baby, 3) a composite pain score (DAN score).

DETAILED DESCRIPTION:
The investigators want to show that the short term autonomic nervous system (ANS) response, after a nociceptive action in the new-born in maternity depends on whether it is preceded by non-nutritive sucking and / or sucrose administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Newborn in maternity unit of the Saint-Etienne University Hospital (France), to receive venipuncture for blood tests or neonatal screening test
* Establishing consent form signed by the holder of parental authority

Exclusion Criteria:

* Children suffering from a disease affecting the central nervous system.
* Children treated with paracetamol oral solution (if cephalohematoma for example) or other analgesics (nalbuphine) or sedative, at the time of registration.
* Newborns impregnated with a prepartum maternal analgesia.

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
High frequency normalized index (HFnu) | From 15 min before the painful care to 15 min after.
  It is a reflect of the RR short term heart rate variability (HRV) in the frequency domain. It is measured with a ECG Holter monitor.

SECONDARY OUTCOMES:
Low frequency (LF and LFnu), | From 15 min before the painful care to 15 min after.
  It is another index of RR heart rate variability (HRV) measured with a ECG Holter monitor.
Scale of hetero-assessment of pain (DAN) | 15 minutes after the painful care
  The DAN scale is specific to acute pain of the newborn
Electro acoustical characteristic of crying newborn : Duration | From 15 min before the painful care to 15 min after.
  An acoustic recording of children's tears will be conducted in parallel with a microphone and dedicated software to study the properties of crying caused by the puncture. Continuous recording begins at least fifteen minutes before the procedure and is kept up to fifteen minutes after the invasive procedure. The child must be quiet. It will be placed in its cocoon to limit environmental stress
Frequency domain | From 15 min before the painful care to 15 min after.
  It is another index of RR heart rate variability (HRV) measured with a ECG Holter monitor.
The time domain (SDNN, SDANN, pNN50). | From 15 min before the painful care to 15 min after.
  It is another index of RR heart rate variability (HRV) measured with a ECG Holter monitor.
LF / HF ratio | From 15 min before the painful care to 15 min after.
  It is another index of RR heart rate variability (HRV) measured with a ECG Holter monitor.
Electro acoustical characteristic of crying newborn : Frequency | From 15 min before the painful care to 15 min after.
  An acoustic recording of children's tears will be conducted in parallel with a microphone and dedicated software to study the properties of crying caused by the puncture. Continuous recording begins at least fifteen minutes before the procedure and is kept up to fifteen minutes after the invasive procedure. The child must be quiet. It will be placed in its cocoon to limit environmental stress
Electro acoustical characteristic of crying newborn : Frequency variations | From 15 min before the painful care to 15 min after.
  An acoustic recording of children's tears will be conducted in parallel with a microphone and dedicated software to study the properties of crying caused by the puncture. Continuous recording begins at least fifteen minutes before the procedure and is kept up to fifteen minutes after the invasive procedure. The child must be quiet. It will be placed in its cocoon to limit environmental stress

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No